CLINICAL TRIAL: NCT02685059
Title: A Randomized Phase II Study to Investigate the Addition of PD-L1 Antibody MEDI4736 to a Taxane-anthracycline Containing Chemotherapy in Triple Negative Breast Cancer (GeparNuevo)
Brief Title: Addition of PD-L1 Antibody MEDI4736 to a Taxane-anthracycline Chemotherapy in Triple Negative Breast Cancer
Acronym: GeparNuevo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: AstraZeneca (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBG89
Record Dates: First submitted 2016-01-14; First posted 2016-02-18 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; Medi4736; Anti PD-L1; Nab-Paclitaxel; Placebo; triple negative
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; 130-nm albumin-bound paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MEDI4736 (Experimental): part 1: MEDI4736 (with half dose as monotherapy for the first two weeks) part 2: MEDI4736 1.5 g total for 20 weeks
  Interventions: Drug: MEDI4736 (Anti PD-L1)
- Placebo (Placebo Comparator): part 1: Placebo (for the first two weeks) part 2: Placebo for 20 weeks
  Interventions: Drug: Placebo
- Taxane (Active Comparator): Nab-Paclitaxel 125 mg/m² weekly for 12 weeks
  Interventions: Drug: nab-Paclitaxel
- Epirubicin (Active Comparator): Epirubicin 90 mg/m² 2-weekly for 8 weeks
  Interventions: Drug: Epirubicin
- Cyclophosphamide (Active Comparator): Cyclophosphamide 600 mg/m² 2-weekly for 8 weeks
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: MEDI4736 (Anti PD-L1) — MEDI4736 1.5g total i.v. every 4 weeks
  As monotherapy for the first two weeks (0.75g absolute) (part 1) followed by:
  MEDI4736 in combination with nab-paclitaxel 125 mg/m² every week for 12 weeks (part 2) followed by
  MEDI4736 in combination with epirubicin 90mg/m² plus cyclophosphamide 600 mg/m² every 2 weeks for 4 cycles (part 3).
  Other Names: Antibody against cell death ligand 1 (PD-L1)
  Arms: MEDI4736
Drug: Placebo — Placebo i.v. every 4 weeks
  As monotherapy for the first two weeks (0.75g absolute) (part 1) followed by:
  Placebo in combination with nab-paclitaxel 125 mg/m² every week for 12 weeks (part 2) followed by
  MEDI4736/Placebo in combination with epirubicin 90mg/m² plus cyclophosphamide 600 mg/m² every 2 weeks for 4 cycles (part 3).
  Arms: Placebo
Drug: nab-Paclitaxel — nab-Paclitaxel 125 mg/m² weekly for 12 weeks
  Other Names: non-solvent based taxane
  Arms: Taxane
Drug: Epirubicin — Epirubicin 90 mg/m² 2-weekly for 8 weeks
  Other Names: Farmorubicin
  Arms: Epirubicin
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m² 2-weekly for 8 weeks
  Other Names: Endoxan
  Arms: Cyclophosphamide

SUMMARY:
To date no targeted agents are available to treat TNBC. Therefore chemotherapy is the only treatment option. TNBC often has a high amount of tumour infiltrating lymphocytes. Stimulating the immune cells of TNBC might therefore be an option for these patients to increase the pathological complete response. pCR is highly correlated with outcome in TNBC.

Therefore the addition of a checkpoint inhibitor in addition to chemotherapy might be an additional option for these patients.

DETAILED DESCRIPTION:
To date no targeted agents are available to treat TNBC. Therefore chemotherapy is the only treatment option. TNBC often has a high amount of tumour infiltrating lymphocytes. Stimulating the immune cells of TNBC might therefore be an option for these patients to increase the pathological complete response. pCR is highly correlated with outcome in TNBC.

Therefore the addition of a checkpoint inhibitor in addition to chemotherapy might be an additional option for these patients.

The primary objective therefore is to compare the pathological complete response (pCR= ypT0 ypN0) rates of neoadjuvant treatment of sequential, nab-Paclitaxel followed by EC +/- the PD-L1 antibody MEDI4736 in patients with early triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for all study according to local regulatory requirements prior to beginning specific protocol procedures.
* Complete baseline documentation must be sent to GBG Forschungs GmbH.
* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration alone is not sufficient. Incisional biopsy is not allowed. In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
* Tumor lesion in the breast or the nodes must be measurable in two dimensions, preferably by sonography. In case of inflammatory disease, the extent of inflammation can be used as measurable lesion.
* Patients must be in the following stages of disease: cT1b - cT4a-d irrespective of nodal involvement.

In patients with multifocal or multicentric breast cancer, the largest lesion should be measured.

* Triple negative disease with centrally confirmed ER negative/PR negative/HER-2 negative, and centrally confirmed Ki-67 value. ER negative is defined as <1% stained cells, PR negative is defined as <10% stained and HER2-negative is defined as either IHC 0/1+ or IHC 2+ and in-situ hybridisation (ISH) of either ratio <2.0 or less than 6 copies of HER2 per tumor cell. Stromal TILs will be evaluated in three groups: low immune infiltrate (0-10% stromal TILs) intermediate immune infiltrate (11-59% stromal TILs), LPBC 60-100% stromal TILs. PD-L1 status and other predefined markers will be prospectively assessed during the study. Formalin-fixed, paraffin-embedded (FFPE) breast tissue from core biopsy has therefore to be sent to the GBG central pathology laboratory prior to randomization.
* Age >=18 years.
* ECOG Performance status 0-1.
* Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 3 months prior to randomization. Results must be above the normal limit of the institution.
* Negative pregnancy test (urine or serum) within 14 days prior to randomization for all women of childbearing potential. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: >=60 years old and no menses for >=1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Complete staging work-up within 3 months prior to randomization. All patients must have had breast imaging by breast ultrasound plus either bilateral mammography or breast MRI (one of those <= 21 days). All patients must have had chest X-ray (PA and lateral), abdominal ultrasound or CT scan or MRI, and bone scan (according to guidelines). In case of positive bone scan, bone X-ray is mandatory. Other tests may be performed as clinically indicated.
* Patients must be available and compliant for central diagnostics, treatment and follow-up.
* Laboratory requirements: Hematology, Hepatic function, Renal Function, Thyroid function

Exclusion Criteria:

* Prior chemotherapy for any malignancy.
* Prior radiation therapy for breast cancer.
* Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization) during study treatment.
* Inadequate general condition (not fit for dose-dense, dose-intensified anthracycline-taxane-targeted agents-based chemotherapy).
* Previous malignant disease being disease-free for less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
* 6. Known or suspected congestive heart failure (>NYHA I) and / or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP >140 / 90 mm Hg under treatment with at maximum two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Bazett's Correction
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* Known history of previous clinical diagnosis of tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving MEDI4736
* Autoimmune disease and conditions (i.e. inflammatory bowel disease)
* History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Pre-existing motor or sensory neuropathy of a severity >= grade 2 by NCI-CTC criteria v 4.0.
* Currently active infection.
* Incomplete wound healing or unhealed bone fracture.
* Definite contraindications for the use of corticosteroids
* Known hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol;
* Concurrent treatment with:
* chronic corticosteroids prior to study entry with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or equivalent corticosteroid.
* other immunosuppressive medication (e.g. low dose MTX)
* sex hormones (including hormonal contraception) prior treatment must be stopped before study entry.
* other experimental drugs or any other anti-cancer therapy.
* Participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including MEDI4736
* Male patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
pathological complete response (pCR= ypT0 ypN0) | 22 weeks
  To compare the pathological complete response (pCR= ypT0 ypN0) rates of neoadjuvant treatment of sequential, nab-Paclitaxel followed by EC +/- the PD-L1 antibody MEDI4736 in patients with early triple negative breast cancer.

SECONDARY OUTCOMES:
pCR rates per arm | 22 weeks
  To assess the pCR rates per arm separately for the stratified subpopulations.
Rates of ypT0/is ypN0 | 22 weeks
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) after treatment in different arms.
Rates of ypT0/is ypN0/+ | 22 weeks
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) after treatment in different arms.
Rates of ypT(any) ypN0 | 22 weeks
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) after treatment in different arms.
Rates of ypT0 ypN0/+ | 22 weeks
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) after treatment in different arms.
Clinical response | 22 weeks
  To assess clinical response rate after taxane in both groups.
Breast conservation rate | 22 weeks
  To determine the breast conservation rate after each treatment.
Toxicity and compliance as measured by number of participants with treatment-related | 22 weeks
  Number of participants with treatment-related adverse events CTCAE v4.0
Molecular markers and gene expression | 22 weeks
  To examine and compare pre-specified molecular markers and gene expression signatures such as tumor infiltrating lymphocytes, PD-1, PD-L1, Ki-67, etc. on core biopsies before chemotherapy, after the window phase and surgical tissue after end of chemotherapy (in %)
Survival | 22 weeks
  To determine loco-regional invasive recurrence free survival (LRRFS), distant-disease-free survival (DDFS), invasive disease-free survival (IDFS), event free survival (EFS per FDA definition) and overall survival (OS) in different arms and according to stratified subpopulations (in months)

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, Prof. Dr., Principal Investigator — GBG Forschungs GmbH
Locations (1):
- Centrum für Hämatologie und Onkologie am Bethanien-Krankenhaus, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Massa C, Karn T, Denkert C, Schneeweiss A, Hanusch C, Blohmer JU, Zahm DM, Jackisch C, van Mackelenbergh M, Thomalla J, Marme F, Huober J, Muller V, Schem C, Mueller A, Stickeler E, Biehl K, Fasching PA, Untch M, Loibl S, Weber K, Seliger B. Differential effect on different immune subsets of neoadjuvant chemotherapy in patients with TNBC. J Immunother Cancer. 2020 Nov;8(2):e001261. doi: 10.1136/jitc-2020-001261. PMID 33199511
- [Derived] Perez-Garcia J, Soberino J, Racca F, Gion M, Stradella A, Cortes J. Atezolizumab in the treatment of metastatic triple-negative breast cancer. Expert Opin Biol Ther. 2020 Sep;20(9):981-989. doi: 10.1080/14712598.2020.1769063. Epub 2020 May 25. PMID 32450725
- [Derived] Loibl S, Untch M, Burchardi N, Huober J, Sinn BV, Blohmer JU, Grischke EM, Furlanetto J, Tesch H, Hanusch C, Engels K, Rezai M, Jackisch C, Schmitt WD, von Minckwitz G, Thomalla J, Kummel S, Rautenberg B, Fasching PA, Weber K, Rhiem K, Denkert C, Schneeweiss A. A randomised phase II study investigating durvalumab in addition to an anthracycline taxane-based neoadjuvant therapy in early triple-negative breast cancer: clinical results and biomarker analysis of GeparNuevo study. Ann Oncol. 2019 Aug 1;30(8):1279-1288. doi: 10.1093/annonc/mdz158. PMID 31095287
- See also: Sponsor study homepage — https://www.gbg.de/de/studien/geparnuevo.php